CLINICAL TRIAL: NCT01580137
Title: Acute Upper Respiratory Tract Infection - When is Bacteria Involved?
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Oulu University Hospital (Other)
Collaborators: Finnish Defense Forces (Other Government); The Central Hospital of Kajaani (Unknown); Huslab, Clinical Microbiology, Virology and Immunology (Unknown); University of Oulu (Other)
Responsible Party: Sponsor
Other Study IDs: Diary number 235/2011
Record Dates: First submitted 2012-04-17; First posted 2012-04-18 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-10

CONDITIONS: Acute Upper Respiratory Tract Infection and Acute Bacterial Rhinosinusitis
Keywords: acute respiratory tract infection; common cold; acute bacterial rhinosinusitis; adult; conscript
MeSH Terms: conditions — Common Cold

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- healthy conscripts: non allergic subjects who have not a history of recurrent rhinosinusitis
- subjects with recurrent rhinosinusitis: subjects who have experienced recurrent rhinosinusitis episodes (3 during the previous 3 years)

SUMMARY:
The purpose of this study is to find out if we can predict the progress of acute upper respiratory tract infection to acute bacterial rhinosinusitis in Finnish conscripts by symptoms, clinical, endoscopic or radiological findings, middle meatal swab samples or nitric oxide measurement.

DETAILED DESCRIPTION:
We will recruit conscripts with upper respiratory tract infection (common cold) during a two month period. We will recruit non-allergic conscripts. These conscripts should either have not had history of recurrent ABR or they should have experienced recurrent acute (ABR) bacterial rhinosinusitis at least 3 times during the last two years (diagnosed by a doctor and at least one time with x-ray or sinus puncture). The recruits will keep a record of their symptoms. They will be examined by a doctor soon after the symptoms have started (2-4 days) and when the symptoms have lasted about 7-10 days. Clinical examination, nasal endoscopy and ultrasonographic examination of the maxillary sinuses are made, middle meatal specimen for bacteria and bacteria-pcr are taken, virus-pcr samples are taken from the nostril and nasopharynx, Nitric oxide-measurements from both nasal cavities are recorded. Cone beam CT of the maxillary and ethmoidal sinuses is made during the first examination, 2-4 days later and during the last examination. If the last CT-scan shows any other radiological signs than mild mucosal oedema in either maxillary sinus, maxillar sinus puncture is made and secretion is aspirated for culture and PCR. Biopsy from the mucosa of nasal cavity (middle meatal area) is taken to examine the cilia and possible bacteria biofilm.

ELIGIBILITY:
Inclusion Criteria:

* Conscript with acute upper respiratory tract infection symptoms (nasal obstruction/decongestion, post nasal drip or nasal secretion) lasted for 2-4 days

Exclusion Criteria:

* Allergy, asthma, nasal polyposis, sinus surgery, autoimmune illness

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Finnish conscripts from the prigade of Kainuu who suffer from acute common cold with nasal symptoms. Consecutive sample. Subjects with known allergies, nasal polyps and prior sinus surgery are excluded.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2012-02; Primary Completion 2012-04 (Actual); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Bacterial maxillary sinusitis | 2 months
  Bacterial maxillary sinusitis defined as positive culture results from the maxillary puncture (either side)

SECONDARY OUTCOMES:
Bacterial sinusitis | 2 months
  positive bacterial pcr results from either maxillary sinus

CONTACTS AND LOCATIONS:
Overall Officials: Petri Koivunen, Dosent, Principal Investigator — Dept of Otolaryngology, University of Oulu, Finland; Timo Koskenkorva, MD, Principal Investigator — Dept of Otolaryngology, University of Oulu, Finland; Mervi Närkiö, MD, Principal Investigator — Finnish Defence Force
Locations (1):
- Finnish Defence Force, Centre for Military Medicine, Kajaani, Kainuu, Finland